CLINICAL TRIAL: NCT06502236
Title: Motor Imagery Ability and Its Relationship With Pain, Functional Status, Neck Awareness and Depression Levels in Individuals With Cervical Discogenic Pain
Brief Title: Motor Imagery Ability and Cervical Discogenic Pain
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, T Dere, Yozgat Bozok University, Hacettepe University
Other Study IDs: MImagery
Record Dates: First submitted 2024-07-07; First posted 2024-07-16 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Motor Imagery; Neck Pain; Disc Herniation; Functional Status
Keywords: Awareness; Endurance; Functional Status; Motor Imagery; Neck; Pain
MeSH Terms: conditions — Neck Pain; Intervertebral Disc Displacement; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control Group: The present study was conducted with individuals aged 18 to 65 years with cervical disc herniation, who were suffered from neck pain lasting for at least 3 months, had a resting pain between 3-7 according to the "Visual Analog Scale" [4], and could follow the instructions of a physiotherapist. All individuals initially diagnosed as cervical disc lesion either one level or multilevel lesions, as diagnosed by the neurologist and confirmed by MRI imaging. The individuals with disk degeneration without cervical disk herniation, cervical stenosis and cervical spondylosis were excluded. In addition, individuals who had a history of spinal tumor or head trauma, had a spinal deformity or congenital malformation, had a cervical instability and cervical artery dysfunction, underwent any cervical surgery in the preceding 6 months, musculoskeletal disorders and neuromuscular diseases in the upper extremity and shoulders.

SUMMARY:
Background: The purpose of the study was to examine the motor imagery ability and its association with pain, functional status, neck awareness and depression levels in individuals with cervical discogenic pain (CDP).

Methods: Sixty individuals aged between 18-65 were included in the study. Demographic data was recorded, pain and disability were evaluated using Visual Analogue Scale (VAS) and Neck Disability Index (NDI), motor imagery ability using Kinesthetic and Visual Imagery Questionnaire-20 (KVIQ-20) and mental chronometry. Grip strength, cervical muscle endurance, upper limbs functionality, neck awareness and depression levels were assessed using hydraulic hand dynamometer, cervical muscle endurance tests, Upper Extremity Functional Index-15 (UEFI-15), Fremantle Neck Awareness Questionnaire (FreNAQ), and Beck Depression Inventory (BDI), respectively.

DETAILED DESCRIPTION:
Motor imagery (MI) is defined as the cognitive representation of a body movement without the actual movement. MI depends on both kinesthetic - which require sensory-motor knowledge- and visual strategies - which require visual knowledge of the movement imagined. Kinesthetic MI is the ability to visualize a movement simulation to perceive its direction, speed, and magnitude. This ability requires the activation of neurocognitive mechanisms that underlie the design and execution of voluntary movement. Visual motor imagery occurs through internal or external visual imagery. Internal visual imagery involves visualizing a movement from ones own perspective, while external visual imagery involves seeing a movement from a third persons perspective. Neuroimaging studies revealed that the parts of the brain activating during MI were similar to those which activate while a movement was actually performed. Therefore, activating joint and muscle receptors by MI may increase corticomotor excitability. Moreover, it was demonstrated that subcortical structures were activated through excitability of presynaptic interneurons by MI, i.e. without activating alpha-motor neurons. Activation through MI ensures continuity of movement and improves the quality of desired movements, playing a key role in enhancing motor function and performance.

Individuals with cervical disc pathologies exhibit a reduced fiber density along the corticospinal tract. Functional magnetic resonance imaging studies have shown increased activation in the primary motor and premotor cortices and a loss of activation in the sensory cortex. These changes are related to the severity of the disc pathology. Besides, it was reported that prolonged compression in the cervical spine might lead to atrophy in the sensorimotor cortex and thalamus, giving rise to a functional reorganization, usually result in maladaptive neuroplasticity. Chronic pain, a common finding in cervical disc pathologies, may affect the perception of painful body parts and MI performance, as well as impaired somatotopic representation. In addition to cortical changes, the gradual processing of stimuli by mirror neurons, which generate motor movements, is considered a significant component of learning by imitation and observation. This process forms an important part of MI and is thought to be impaired in individuals with chronic pain. They highlighted that evaluating the MI ability of an individual with chronic neck pain was important for revealing the mental imagery performance.

In individuals with chronic neck pain, it was revealed that the severity of pain and the functional and psychosocial problems caused by the pain, were related to executive functions and working memory. They discovered that MI depends on executive functions. Interference tasks significantly affect the timing of MI. Therefore, it is believed that pain-related symptoms will also negatively impact MI skills. In the literature, studies have demonstrated positive effects of MI training on pain, disability, and fear of movement in individuals with chronic pain. However, it is suggested that factors related to MI ability should be further investigated. Therefore, the purpose of the study was to examine the relationships between MI ability and pain, functional status, neck awareness and depression levels in individuals with cervical discogenic pain (CDP).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years with cervical disc herniation, who were suffered from neck pain lasting for at least 3 months,
* Had a resting pain between 3-7 according to the Visual Analog Scale;
* Could follow the instructions of a physiotherapist.

Exclusion Criteria:

* The individuals with disk degeneration without cervical disk herniation, cervical stenosis and cervical spondylosis were excluded.
* In addition, individuals who had a history of spinal tumor or head trauma, had a spinal deformity or congenital malformation, had a cervical instability and cervical artery dysfunction, underwent any cervical surgery in the preceding 6 months, musculoskeletal disorders and neuromuscular diseases in the upper extremity and shoulders (rotator cuff tear, very severe myofascial pain syndrome, cervical facet joint pain, carpal tunnel disease, etc.)
* Who were not able to follow the instructions of the therapist were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The present study was conducted with individuals aged 18 to 65 years with cervical disc herniation, who were suffered from neck pain lasting for at least 3 months, had a resting pain between 3-7 according to the Visual Analog Scale and could follow the instructions of a physiotherapist. All individuals initially diagnosed as cervical disc lesion either one level or multilevel lesions, as diagnosed by the neurologist and confirmed by MRI imaging. The individuals with disk degeneration without cervical disk herniation, cervical stenosis and cervical spondylosis were excluded.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain Severity | February 2024
  The 10-cm Visual Analogue Scale (VAS) developed by Price et al., and The Neck Disability Index (NDI) developed by Vernon et al. were used to evaluate the pain severity and the disability related to neck. On the 10-cm VAS, the first notch is marked 0, and the last notch is marked 10. Zero means no pain, whereas 10 means the most severe pain.
Assessment of Neck Disability | February 2024
  The Neck Disability Index (NDI) developed by Vernon et al. was used to evaluate the disability caused by chronic neck pain. Validated for reliability in Turkish by Aslan et al., the questionnaire is made up of 10 questions questioning the impact of neck pain on daily activities including personal care, concentration, working, driving and sleeping. Each question is rated between 0 and 5 with the maximum score being 50. 0 to 4 points means no disability, 5 to 14 points means mild disability, 14 to 24 points means moderate disability, 25 to 34 points means serious disability, 35 and above means complete disability, and 50 points means full disability .
Assessment of Motor Imagery Ability | February 2024
  MI skills of the participants were evaluated with the Kinesthetic and Visual Imagery Questionnaire-20 (KVIQ-20) developed to determine the extent to which individuals can visualize and sense an imagined movement. Validated for reliability in Turkish by Dilek et al., the questionnaire included 20 movements measuring 10 visual and 10 kinesthetic imagery skills. To perform the assessment, first, the physiotherapist showed the required movement on their own body, and then asked the participant to repeat that movement physically once. Then the participants were asked to imagine the movement and rate the movement for how much it was felt based on its visual clarity. The overall score included the sum of separate scores of kinesthetic imagery skill and visual imagery skill and ranged between 20 and 100. Higher scores indicated higher clarity and intensity of sensation

SECONDARY OUTCOMES:
Assessment of Grip Strength | February 2024
  The grip strength of the individuals was evaluated by a hydraulic hand dynamometer (Baseline lite Hydraulic Hand Dynamometer, Fabrication Enterprises, NY, USA), and the result was noted in kilograms.
Assessment of Muscular Endurance-Flexor | February 2024
  The endurance of the neck flexors of the participants were evaluated in the supine hooked position with the head placed 6 cm high. After taking the height below the head, the maximum time maintaining this position was noted in seconds. The 5-degree change in a goniometer following the vertical angle of the mandible was determined as the criterion for terminating the test
Assessment of Muscular Endurance-Extensor | February 2024
  The neck extensor muscle endurance of the participants was evaluated by attaching a 2-kg weight using a 10-cm velcro at the C6 level in a prone position with the hands placed to both sides. The maximum duration of holding head in this position was recorded in seconds.
Assessment of Muscular Endurance-Deep Flexor | February 2024
  Cervical deep flexor muscle endurance of the participants was evaluated in supine hooked position with the hands placed on the abdomen and the chin pulled in. The maximum time the participant could raise and hold their head about 2.5 cm high was noted.
Assessment of Neck Awareness | February 2024
  Neck awareness levels of the participants were evaluated by the Fremantle Neck Awareness Questionnaire (FreNAQ). Validated for reliability in Turkish by Onan et al., the questionnaire is made up of 9 questions measuring neck pain, attention and proprioceptive awareness. Each question is rated between 0 (Never/I never feel this way) and 4 (I always or usually feel this way). The overall score ranges between 0 to 36 with a higher score indicating poor neck awareness .
Assessment of Upper Extremity Functionality | February 2024
  Upper extremity functionality of the participants was evaluated with the Upper Extremity Functional Index-15 (UEFI-15). Validated for reliability in Turkish by Aytar et al., the questionnaire includes 15 different activities that are frequently carried out in daily life. Individuals are asked to rate each activity by the level of difficulty performing it on a scoring system ranged from 0 (extremely difficult) to 4 (no difficulty). The overall score ranges between 0-100. Lower scores indicate poor upper extremity functionality
Assessment of Depression Level | February 2024
  Depression levels of the participants were evaluated by the Beck Depression Inventory (BDI). The participants were asked to answer 21 questions assessing depressive behaviors, rating them from 0 to 3. Validated for reliability in Turkish by Kapci et al., the questionnaire has an overall score range of 0 to 63 points. 0 to 12 points means minimal depression; 13 to 18 points, mild depression; 19 to 28 points, moderate depression; and 29 to 63 points, serious depression.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Dere, MSc, Principal Investigator — Yozgat Bozok University
Locations (1):
- Sarıkaya Physical Therapy and Rehabilitation High School, Yozgat, Sarıkaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] undefined
- [Result] Wang C, Laiwalla A, Salamon N, Ellingson BM, Holly LT. Compensatory brainstem functional and structural connectivity in patients with degenerative cervical myelopathy by probabilistic tractography and functional MRI. Brain Res. 2020 Dec 15;1749:147129. doi: 10.1016/j.brainres.2020.147129. Epub 2020 Sep 17. PMID 32950486
- [Result] Suica Z, Platteau-Waldmeier P, Koppel S, Schmidt-Trucksaess A, Ettlin T, Schuster-Amft C. Motor imagery ability assessments in four disciplines: protocol for a systematic review. BMJ Open. 2018 Dec 14;8(12):e023439. doi: 10.1136/bmjopen-2018-023439. PMID 30552265
- [Result] Javdaneh N, Molayei F, Kamranifraz N. Effect of adding motor imagery training to neck stabilization exercises on pain, disability and kinesiophobia in patients with chronic neck pain. Complement Ther Clin Pract. 2021 Feb;42:101263. doi: 10.1016/j.ctcp.2020.101263. Epub 2020 Nov 19. PMID 33276225
- [Result] Lebon F, Guillot A, Collet C. Increased muscle activation following motor imagery during the rehabilitation of the anterior cruciate ligament. Appl Psychophysiol Biofeedback. 2012 Mar;37(1):45-51. doi: 10.1007/s10484-011-9175-9. PMID 22127572
- [Derived] Dere T, Yurdakul G, Bugra Kilinc S, Alemdaroglu-Gurbuz I. Association Between Motor Imagery Ability and Pain, Functional Status, Neck Awareness, and Depression in Individuals with Chronic Neck Pain. Altern Ther Health Med. 2025 Mar;31(2):23-29. PMID 39715569